CLINICAL TRIAL: NCT03630055
Title: Rivaroxaban Post-Transradial Access for the Prevention of Radial Artery Occlusion
Acronym: CAPITAL-RAPTOR
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20180319; NCT05399277 (obsolete NCT alias)
Record Dates: First submitted 2018-07-19; First posted 2018-08-14 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2024-07

CONDITIONS: Radial Artery Occlusion
Keywords: Direct oral anticoagulants; Transradial access; Percutaneous coronary intervention
MeSH Terms: conditions — Arterial Occlusive Diseases | interventions — Rivaroxaban; Tablets

STUDY DESIGN:
Intervention Model Description: Eligible patients will undergo a 1:1 randomization using a computer-generated randomization sequence to either receive a direct oral anticoagulant (i.e. rivaroxaban 15mg oral daily) for 7 days or to the standard of care arm (i.e. no rivaroxaban)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rivaroxaban (Experimental): Participants will receive rivaroxaban 15mg tablet to be taken orally once daily for 7 days. Follow up will be within 30 days where participants will undergo a Doppler ultrasound to assess for radial artery patency/occlusion.
  Interventions: Drug: Rivaroxaban 15 MG Oral Tablet [Xarelto]
- Standard of Care (No Intervention): Participants will not receive any anticoagulation. Follow up will be within 30 days where participants will undergo a Doppler ultrasound to assess for radial artery patency/occlusion.

INTERVENTIONS:
Drug: Rivaroxaban 15 MG Oral Tablet [Xarelto] — Patients will receive rivaroxaban 15mg orally daily for 7 days following transradial access.
  Other Names: Xarelto
  Arms: Rivaroxaban

SUMMARY:
Coronary angiography is performed to evaluate for obstructive coronary artery disease. This is commonly performed via the transfemoral or transradial approach with the latter increasing in frequency. One of the most common complications of transradial access is radial artery occlusion occurring in ~5% of patients which prohibits the use of the radial artery in the future. There is evidence to support the use of intraprocedural anticoagulation to mitigate the risk of radial artery occlusion however the role of post-procedural anticoagulation has not been previously evaluated. Rivaroxaban is a direct oral anticoagulant (DOAC) with a safety profile superior to that of vitamin K antagonists. Given the safety profile, ease of use, and feasibility of DOAC therapy, our study will endeavor to evaluate the use of rivaroxaban 15mg orally once daily for 7 days after transradial access and the impact this has on the rate of radial artery occlusion.

DETAILED DESCRIPTION:
Assessment of the coronary artery anatomy is commonly performed by coronary angiography (CA), which is the gold standard for evaluation of obstructive coronary artery disease (CAD). Coronary revascularization, opening of obstructed vessels, is most commonly performed by percutaneous coronary intervention (PCI) in patients with obstructive CAD. Traditionally, PCI is performed with implantation of one or more permanent metallic stents which act as a scaffold for arterial recoil and, in the case of drug eluting stents (DES), provide a platform for delivery of anti-proliferative agents. The transradial access (TRA) has rapidly emerged as the preferred vascular access site for CA and PCI with more than 50% of all coronary angiograms being performed via this approach.

There are several advantages to TRA for angiography including rapid hemostasis, early ambulation after the procedure thereby improving patient comfort and experience, and a decrease in the length of hospital stay. There is also a reported reduction in all-cause mortality, major adverse cardiovascular events, major bleeding, and vascular complications with TRA as compared to transfemoral access. However, radial artery occlusion (RAO) remains an important complication of this procedure as it precludes the reuse of this artery for future transradial approaches as well as the use of the vessel as a conduit for coronary artery bypass grafting.

Reports of RAO post-TRA has varied in the literature from ~4-10% in observational and randomized trials. In the largest systematic review published to date, the overall rate of RAO was 5.2% amongst the 46,631 subjects across 92 studies between 1989 and 2016. This systematic review also noted that the rate of early (i.e. <7 days) vs. late (i.e. >7 days) RAO was significantly higher which is suggestive of late recanalization in some patients. The factors which affect recanalization are not clear however standard of care involves administration of heparin during the procedure and patent hemostasis following the procedure. Patent hemostasis is performed by applying a delicate balance of pressure to prevent bleeding but not to the point of completely occlude the blood vessel and cessation of blood flow distally.

Numerous trials have explored the role of anticoagulation during angiography to reduce RAO and a recently published systematic review and meta-analysis demonstrated more intensive anticoagulation is protective. Indeed, this remains an active area of research with numerous ongoing trials evaluating the effect of intensive or higher dose anticoagulation during the procedure for prevention of RAO. Additionally, there were higher rates of RAO with diagnostic angiography as opposed to PCI purportedly as the latter involves higher doses of anticoagulation.

Direct oral anticoagulant (DOAC) therapy has provided a safer alternative with an improved bleeding profile over vitamin K antagonist anticoagulation therapy. The use of DOACs in cardiovascular medicine ranges from various conditions including stroke prevention in atrial fibrillation7-12 to venous thromboembolism13-16 to stable cardiovascular disease.

While intraprocedural anticoagulation has been studied extensively, a course of anticoagulation therapy post-TRA has not been studied. Given the safety profile, ease of use, and feasibility of DOAC therapy, our study will endeavor to evaluate the use of rivaroxaban 15mg orally once daily for 7 days after transradial access and the impact this has on the rate of RAO. Should this study prove to be positive, this could impact our routine standard of care with respect to having a strategy which could reduce the rate of this complication thereby preserving the radial artery for future access and/or as a conduit for coronary artery bypass grafting.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent
2. Age ≥ 18 years
3. Diagnostic coronary angiography or percutaneous coronary intervention via the transradial approach

Exclusion Criteria:

1. Presence of a palpable hematoma or clinical concern of hemostasis at the transradial access site
2. Access or attempted access at a second site - including contralateral radial artery, brachial, or femoral artery or vein
3. Planned staged procedure, CABG or noncardiac surgery within 30 days
4. Contraindication or high risk of bleeding with anticoagulation

   1. bleeding requiring medical attention in the previous 6 months
   2. thrombocytopenia (platelets<50 x 109/L)
   3. prior intracranial hemorrhage
   4. use of IIb/IIIa during percutaneous coronary intervention
   5. administration of thrombolytic therapy in the preceding 24 hours
   6. use of non-steroidal anti-inflammatory medications
   7. ischemic stroke or transient ischemic attack diagnosed in the last 3 months
5. Cardiogenic shock
6. Ventricular arrhythmias refractory to treatment
7. Liver dysfunction (Child-Pugh class B or C)
8. Unexplained anemia with a Hgb below 100 g/L
9. History of medication noncompliance or risk factor for noncompliance
10. Active malignancy
11. Allergy to rivaroxaban
12. Another indication for anticoagulation
13. CYP3A4 and P-glycoprotein inhibitor use
14. Life expectancy <30 days
15. Women capable of pregnancy not on birth control
16. Chronic kidney disease with creatinine clearance of less than 30mL/min
17. History of antiphosphopholipid antibody syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2018-10-03 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy outcome - rate of radial artery occlusion | 30 days
  Presence of radial artery occlusion at 30 days post-transradial access as determined by Doppler ultrasound assessment of the participant's radial artery in the wrist.
Primary safety outcome - International Society on Thrombosis and Haemostasis definition of major bleeding | 30 days
  Bleeding as defined by the International Society on Thrombosis and Haemostasis at 30 days.

SECONDARY OUTCOMES:
All cause mortality | 30 days
  Death from any cause as determined by the treating physician
Stroke (ischemic or uncertain) | 30 days
  Stroke (ischemic or uncertain) as defined by a treating neurologist
Stroke (hemorrhagic) | 30 days
  Stroke (hemorrhagic) as defined by a treating neurologist
Fatal bleeding | 30 days
  Bleeding resulting in death as defined by treating physician
Symptomatic bleeding in a critical area or organ | 30 days
  Intracranial, intraspinal, intraocular, retroperitoneal, intra-articular or pericardial bleeding or intramuscular bleeding with compartment syndrome
Bleeding requiring medical attention | 30 days
  Any bleeding that requires participant to seek medical attention
GUSTO bleeding criteria | 30 days
  Bleeding as defined by the Global Utilization Of Streptokinase And Tpa For Occluded Arteries (GUSTO) criteria
TIMI bleeding criteria | 30 days
  Bleeding as defined by the Thrombolysis in Myocardial Infarction (TIMI) criteria
BARC bleeding criteria | 30 days
  Bleeding as defined by the Bleeding Academic Research Consortium (BARC) criteria
Myocardial infarction | 30 days
  Myocardial infarction as defined by the third universal definition of myocardial infarction.
Stent thrombosis | 30 days
  Stent thrombosis as determined by the academic research consortium criteria.

CONTACTS AND LOCATIONS:
Locations (3):
- Mayo Clinic, Rochester, Minnesota, United States
- Canada (2):
  - Kingston Health Sciences Center, Kingston, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario

REFERENCES:
- [Background] Simard T, Hibbert B, Ramirez FD, Froeschl M, Chen YX, O'Brien ER. The evolution of coronary stents: a brief review. Can J Cardiol. 2014 Jan;30(1):35-45. doi: 10.1016/j.cjca.2013.09.012. Epub 2013 Nov 25. PMID 24286961
- [Background] Bertrand OF, Rao SV, Pancholy S, Jolly SS, Rodes-Cabau J, Larose E, Costerousse O, Hamon M, Mann T. Transradial approach for coronary angiography and interventions: results of the first international transradial practice survey. JACC Cardiovasc Interv. 2010 Oct;3(10):1022-31. doi: 10.1016/j.jcin.2010.07.013. PMID 20965460
- [Background] Schussler JM, Vasudevan A, von Bose LJ, Won JI, McCullough PA. Comparative Efficacy of Transradial Versus Transfemoral Approach for Coronary Angiography and Percutaneous Coronary Intervention. Am J Cardiol. 2016 Aug 15;118(4):482-8. doi: 10.1016/j.amjcard.2016.05.038. Epub 2016 May 29. PMID 27378143
- [Background] Ferrante G, Rao SV, Juni P, Da Costa BR, Reimers B, Condorelli G, Anzuini A, Jolly SS, Bertrand OF, Krucoff MW, Windecker S, Valgimigli M. Radial Versus Femoral Access for Coronary Interventions Across the Entire Spectrum of Patients With Coronary Artery Disease: A Meta-Analysis of Randomized Trials. JACC Cardiovasc Interv. 2016 Jul 25;9(14):1419-34. doi: 10.1016/j.jcin.2016.04.014. Epub 2016 Jun 29. PMID 27372195
- [Background] Hahalis G, Aznaouridis K, Tsigkas G, Davlouros P, Xanthopoulou I, Koutsogiannis N, Koniari I, Leopoulou M, Costerousse O, Tousoulis D, Bertrand OF. Radial Artery and Ulnar Artery Occlusions Following Coronary Procedures and the Impact of Anticoagulation: ARTEMIS (Radial and Ulnar ARTEry Occlusion Meta-AnalysIS) Systematic Review and Meta-Analysis. J Am Heart Assoc. 2017 Aug 23;6(8):e005430. doi: 10.1161/JAHA.116.005430. PMID 28838915
- [Background] Pancholy S, Coppola J, Patel T, Roke-Thomas M. Prevention of radial artery occlusion-patent hemostasis evaluation trial (PROPHET study): a randomized comparison of traditional versus patency documented hemostasis after transradial catheterization. Catheter Cardiovasc Interv. 2008 Sep 1;72(3):335-340. doi: 10.1002/ccd.21639. PMID 18726956
- [Background] Gibson CM, Mehran R, Bode C, Halperin J, Verheugt FW, Wildgoose P, Birmingham M, Ianus J, Burton P, van Eickels M, Korjian S, Daaboul Y, Lip GY, Cohen M, Husted S, Peterson ED, Fox KA. Prevention of Bleeding in Patients with Atrial Fibrillation Undergoing PCI. N Engl J Med. 2016 Dec 22;375(25):2423-2434. doi: 10.1056/NEJMoa1611594. Epub 2016 Nov 14. PMID 27959713
- [Background] Patel MR, Mahaffey KW, Garg J, Pan G, Singer DE, Hacke W, Breithardt G, Halperin JL, Hankey GJ, Piccini JP, Becker RC, Nessel CC, Paolini JF, Berkowitz SD, Fox KA, Califf RM; ROCKET AF Investigators. Rivaroxaban versus warfarin in nonvalvular atrial fibrillation. N Engl J Med. 2011 Sep 8;365(10):883-91. doi: 10.1056/NEJMoa1009638. Epub 2011 Aug 10. PMID 21830957
- [Background] EINSTEIN-PE Investigators; Buller HR, Prins MH, Lensin AW, Decousus H, Jacobson BF, Minar E, Chlumsky J, Verhamme P, Wells P, Agnelli G, Cohen A, Berkowitz SD, Bounameaux H, Davidson BL, Misselwitz F, Gallus AS, Raskob GE, Schellong S, Segers A. Oral rivaroxaban for the treatment of symptomatic pulmonary embolism. N Engl J Med. 2012 Apr 5;366(14):1287-97. doi: 10.1056/NEJMoa1113572. Epub 2012 Mar 26. PMID 22449293
- [Background] Eikelboom JW, Connolly SJ, Bosch J, Dagenais GR, Hart RG, Shestakovska O, Diaz R, Alings M, Lonn EM, Anand SS, Widimsky P, Hori M, Avezum A, Piegas LS, Branch KRH, Probstfield J, Bhatt DL, Zhu J, Liang Y, Maggioni AP, Lopez-Jaramillo P, O'Donnell M, Kakkar AK, Fox KAA, Parkhomenko AN, Ertl G, Stork S, Keltai M, Ryden L, Pogosova N, Dans AL, Lanas F, Commerford PJ, Torp-Pedersen C, Guzik TJ, Verhamme PB, Vinereanu D, Kim JH, Tonkin AM, Lewis BS, Felix C, Yusoff K, Steg PG, Metsarinne KP, Cook Bruns N, Misselwitz F, Chen E, Leong D, Yusuf S; COMPASS Investigators. Rivaroxaban with or without Aspirin in Stable Cardiovascular Disease. N Engl J Med. 2017 Oct 5;377(14):1319-1330. doi: 10.1056/NEJMoa1709118. Epub 2017 Aug 27. PMID 28844192
- [Background] Habib J, Baetz L, Satiani B. Assessment of collateral circulation to the hand prior to radial artery harvest. Vasc Med. 2012 Oct;17(5):352-61. doi: 10.1177/1358863X12451514. Epub 2012 Jul 19. PMID 22814998
- [Background] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242
- [Background] Sabatine MS, Morrow DA, Giugliano RP, Burton PB, Murphy SA, McCabe CH, Gibson CM, Braunwald E. Association of hemoglobin levels with clinical outcomes in acute coronary syndromes. Circulation. 2005 Apr 26;111(16):2042-9. doi: 10.1161/01.CIR.0000162477.70955.5F. Epub 2005 Apr 11. PMID 15824203
- [Background] Rao SV, O'Grady K, Pieper KS, Granger CB, Newby LK, Van de Werf F, Mahaffey KW, Califf RM, Harrington RA. Impact of bleeding severity on clinical outcomes among patients with acute coronary syndromes. Am J Cardiol. 2005 Nov 1;96(9):1200-6. doi: 10.1016/j.amjcard.2005.06.056. Epub 2005 Sep 12. PMID 16253582
- [Background] Schulman S, Kearon C; Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medicinal products in non-surgical patients. J Thromb Haemost. 2005 Apr;3(4):692-4. doi: 10.1111/j.1538-7836.2005.01204.x. PMID 15842354
- [Background] Thygesen K, Alpert JS, Jaffe AS, Simoons ML, Chaitman BR, White HD; Writing Group on behalf of the Joint ESC/ACCF/AHA/WHF Task Force for the Universal Definition of Myocardial Infarction. Third universal definition of myocardial infarction. Glob Heart. 2012 Dec;7(4):275-95. doi: 10.1016/j.gheart.2012.08.001. Epub 2012 Sep 26. No abstract available. PMID 25689940
- [Background] Cutlip DE, Windecker S, Mehran R, Boam A, Cohen DJ, van Es GA, Steg PG, Morel MA, Mauri L, Vranckx P, McFadden E, Lansky A, Hamon M, Krucoff MW, Serruys PW; Academic Research Consortium. Clinical end points in coronary stent trials: a case for standardized definitions. Circulation. 2007 May 1;115(17):2344-51. doi: 10.1161/CIRCULATIONAHA.106.685313. PMID 17470709
- [Derived] Di Santo P, Abdel-Razek O, Jung R, Parlow S, Poulin A, Bernick J, Morgan B, Robinson L, Feagan H, Wade J, Goh CY, Singh K, Froeschl M, Labinaz M, Fergusson DA, Coyle D, Kyeremanteng K, Abunassar J, Wells GA, Simard T, Hibbert B. Rationale and Design of the Rivaroxaban Post-Transradial Access for the Prevention of Radial Artery Occlusion Trial (CAPITAL-RAPTOR). BMJ Open. 2023 May 12;13(5):e070720. doi: 10.1136/bmjopen-2022-070720. PMID 37173116